CLINICAL TRIAL: NCT07083323
Title: A Multicenter, Open-label Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Clinical Efficacy of HY05350 for Injection in Patients With MSLN-positive Advanced Solid Tumors
Brief Title: A Phase I/II Study of HY05350 in Mesothelin(MSLN)-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HY0005-101
Record Dates: First submitted 2025-07-06; First posted 2025-07-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1, the single-agent dose escalation of HY05350 for injection. (Experimental)
  Interventions: Drug: HY05350 for injection
- Part 2, dose expansion. The recommended dose will be established from the Dose Escalation part. (Experimental)
  Interventions: Drug: HY05350 for injection

INTERVENTIONS:
Drug: HY05350 for injection — HY05350 should be administered intravenously at planned dosage, once a week, once every two weeks, or once every three weeks, until disease progression or intolerable toxicity occurs.
  Arms: Part 1, the single-agent dose escalation of HY05350 for injection.
Drug: HY05350 for injection — HY05350 should be administered intravenously at recommended dose, once a week, once every two weeks, or once every three weeks, until disease progression or intolerable toxicity occurs.
  Arms: Part 2, dose expansion. The recommended dose will be established from the Dose Escalation part.

SUMMARY:
This is a multicenter, open-label Phase I/II clinical study to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary clinical efficacy of HY05350 for injection in patients with MSLN-positive advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open-label phase I/II clinical trial divided into two parts: dose escalation part (Part 1) and dose expansion part (Part 2). The main objectives of the first part are to evaluate the safety and tolerability of HY05350 for injection as monotherapy in patients with mesothelin-positive advanced solid tumors, and to explore the Maximum Tolerated Dose (MTD) and determine the Recommended Phase 2 Dose (RP2D) or the recommended dose for subsequent clinical studies. The main objective of the second part is to evaluate the anti-tumor efficacy of HY05350 for injection. The study includes patients with cytologically or pathologically confirmed advanced solid tumors who have failed standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤75 years at the time of signing the informed consent form, regardless of gender.
2. Investigator-assessed expected survival period ≥3 months.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
4. Patients with cytologically or pathologically confirmed advanced solid tumors who have failed standard treatment.
5. Subjects enrolled in the dose escalation stage must have evaluable tumor lesions, and subjects enrolled in the dose expansion stage must have at least one measurable tumor lesion (based on RECIST 1.1).
6. Participant must have adequate main organ function.
7. Agree to provide archived pathological tissues or fresh biopsy tumor tissues for detection of related markers such as MSLN and Programmed cell death ligand 1 (PD-L1) expression levels, and MSLN expression is positive.
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first drug administration, and be willing to use effective contraceptive methods to prevent pregnancy and have no plans to donate eggs during the study period and for 6 months after the last drug administration. Male subjects must agree to have no plans to donate sperm and use effective contraceptive methods during the study period and for 6 months after the last drug administration. Postmenopausal women must have been amenorrheic for at least 12 months to be considered non-childbearing.

Exclusion Criteria:

1. Received radiotherapy, chemotherapy, endocrine therapy, biological therapy, immunotherapy and other anti-tumor therapies within 4 weeks before the first drug administration.
2. Received other investigational drugs or participated in interventional medical device studies within 4 weeks before the first drug administration.
3. Had received or planned to receive live/attenuated vaccines or mRNA vaccines within 4 weeks before screening.
4. Pregnant or lactating women.
5. Subjects with adverse events caused by previous anti-tumor therapy that remained > Grade 1 (based on CTCAE 5.0) before the first drug administration.
6. Subjects with a history of ≥ Grade 3 immune-related adverse events or who discontinued immunotherapy due to irAE of any grade.
7. Subjects with primary central nervous system (CNS) tumors, symptomatic CNS metastases, meningeal metastases, or a history of epilepsy are excluded.
8. Subjects who underwent major surgery on vital organs (excluding biopsy) within 4 weeks before the first drug administration, experienced significant trauma, or require major elective surgery during the trial.
9. Subjects with a history of tissue or organ transplantation.
10. Subjects who had severe infections within 4 weeks before the first drug administration.
11. Positive human immunodeficiency virus test.
12. Active hepatitis B, untreated chronic hepatitis B, or chronic hepatitis B that is treated but uncontrolled.
13. Subjects with active Hepatitis C virus(HCV) infection;
14. Positive treponema pallidum antibody and confirmed positive by diagnostic test;
15. Subjects with untreated or ongoing tuberculosis.
16. Known severe allergic history, or known allergic reactions to macromolecular protein preparations/antibodies or any component of the investigational drug.
17. History of active autoimmune diseases or a history of autoimmune diseases with potential for recurrence.
18. Subjects who received systemic glucocorticoids or other immunosuppressants within 14 days before the first drug administration.
19. History of non-infectious pneumonia requiring glucocorticoid treatment or current interstitial lung disease.
20. History of severe cardiovascular and cerebrovascular diseases.
21. Subjects with thrombosis or bleeding risk.
22. Known history of psychoactive substance abuse or drug use that is considered to affect study compliance.
23. Except for the tumor enrolled in the study, subjects with other active malignant tumors within 1 year before the first drug administration.
24. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage.
25. Subjects deemed unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1, the occurrence of dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days).
  Measure Description: DLT will be defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or American Society for Transplantation and Cellular Therapy (ASTCT) criteria for Cytokine Release Syndrome (CRS).
Part 1, Incidence of Treatment-Emergent Adverse Events (TEAE) | Up to 2 years.
  Measure Description: Incidence and severity of TEAE according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Part 2, Objective Response Rate (ORR) | Up to 2 years.
  Measure Description: The proportion of participants who have a Complete Response (CR) or a Partial Response (PR) based on Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1.

SECONDARY OUTCOMES:
Part 1, Peak Plasma Concentration (Cmax) | At the end of Cycle 3 (each cycle is 28 days).
  Measure Description: Maximum concentration observed from the pharmacokinetic profile
Part 1, Area under the plasma concentration versus time curve (AUC) | At the end of Cycle 3 (each cycle is 28 days).
  Measure Description: Area under the concentration versus time curve calculated using the trapezoidal method.
Part 1, Assessment of Anti-drug Antibody (ADA) | Up to 2 years.
  Measure Description: Incidence, duration, titer of serum anti-HY05350 antibody (ADA)
Part 1, Objective Response Rate (ORR) | Up to 2 years.
  Measure Description: Proportion of participants who have a complete response (CR) or a partial response (PR) determined by Investigator per the Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1.
Part 2, Duration Of Response (DOR) | Up to 2 years.
  Measure Description: Duration Of Response (DOR) is defined as the time from the measurement criteria are first met for complete response (CR) /partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease.
Part 2, Incidence of Treatment-Emergent Adverse Events (TEAE) | Up to 2 years.
  Measure Description: Incidence and severity of TEAE according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Part 2, Peak Plasma Concentration (Cmax) | At the end of Cycle 3 (each cycle is 28 days).
  Measure Description: Maximum concentration observed from the pharmacokinetic profile.
Part 2, Assessment of Anti-drug Antibody (ADA) | Up to 2 years.
  Measure Description: Incidence, duration, titer of serum anti-HY05350 antibody (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wan, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No